CLINICAL TRIAL: NCT05952167
Title: Evaluation of the Impact of Tractions vs. Placebo Tractions in Patients With Cervical Radiculopathy, Randomised Controlled Trial in a Single-blind Study
Brief Title: Evaluation of the Impact of Tractions vs. Placebo Tractions in Patients With Cervical Radiculopathy
Acronym: TracCerv2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHD 22_0054
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Radiculopathy; Cervical
Keywords: Cervical traction; Cervical radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo mechanical cervical traction (Placebo Comparator)
  Interventions: Other: Intensive cervical traction protocol - placebo
- Mechanical cervical traction (Experimental)
  Interventions: Other: Intensive cervical traction protocol

INTERVENTIONS:
Other: Intensive cervical traction protocol — 2x/day over 5 weekdays A minimum of 8 pull-ups over 5 consecutive days is expected.
  Arms: Mechanical cervical traction
Other: Intensive cervical traction protocol - placebo — 2x/day over 5 weekdays A minimum of 8 pull-ups over 5 consecutive days is expected.
  Arms: Placebo mechanical cervical traction

SUMMARY:
Cervical radiculopathy is a common disease related to compression of the nerve roots of the spine (prevalence: 3.5/1000). Dysfunction and pain are the main repercussions and can lead to time off work and high costs in terms of treatment.

Second-line surgical treatments appear to be less effective and present risks of side effects. In the first instance, treatments are conservative and include medication but above all physiotherapy with manual therapy, muscle exercises and cervical traction. These cervical tractions performed by a physiotherapist require little equipment and are inexpensive compared with the surgical alternative. They involve stretching the cervical spine and soft tissues to open the intervertebral foramen and mobilise the facet joints.

Several authors have written summaries of their interest. Thoomes reports two studies and describes an absence of effect. In a meta-analysis, Romeo et al. added three more recent studies to the previous review and concluded that traction is effective, highlighting an "effect-dose" relationship. These recent results therefore seem to reverse the recommendations made barely two years later. Nevertheless, almost all the studies compared "manual therapy + exercises" with "manual therapy + exercises + cervical traction". Only Young et al. tested "manual therapy + exercises + cervical traction at an effective weight" compared to "manual therapy + exercises + cervical traction placebo at an ineffective weight". The study did not reveal any difference between the groups. However, several limitations appear in this study when comparing the protocol to studies that have shown efficacy. The main limitation is the low intensity (i.e. protocol with fewer sessions and longer duration). These clinical limitations may explain the lack of evidence of a positive outcome. Following on from a preliminary study evaluating an intensive cervical traction protocol over five days, and in order to discern the effect specific to the treatment (specific effect) and the effect independent of the nature of the treatment (contextual effect), the investigators wish to evaluate the impact of this intensive protocol by comparing it with placebo traction.

In current practice, treatment varies between establishments. The paucity of studies on cervical traction in radiculopathy has resulted in routine use being guided by habit rather than evidence. It remains a clinical question which raises a major issue requiring a robust experimental design. Ultimately, this study follows on from a preliminary study and is part of a comprehensive research project aimed at proposing new recommendations for the use of traction in patients suffering from cervical radiculopathy. The investigators are investigating the impact of an intensive traction vs. placebo traction protocol in patients with cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18
* Neck Disability Index ≥ 15/50
* Presence of at least three of the four signs clinically validating the presence of cervical radiculopathy (Wainner et al. 2003)

  * a) upper limb nerve tension test A (ULNT1a): positive,
  * b) amplitude of cervical rotation on the side concerned: < 60°,
  * c) positive cervical distraction test: relief
  * d) positive Spurling test: reproduction of symptoms.
* Cervical radiculopathy diagnosed 3 to 24 months previously
* Absence of cervical traction in the 5 years prior to inclusion
* MRI or CT scan performed prior to hospitalisation in relation to current pathology
* Patient able to understand the protocol and having given oral informed consent to take part in the research.
* Patient affiliated to the social security system or entitled beneficiary.

Exclusion Criteria:

* Patients with vertebral artery pathology at the time of inclusion
* Patients with myelopathy, cervical cancer, cervical fracture, cervical dislocation, cervical spondylolisthesis, spinal infection, symptomatic cervical pain without radiculopathy and/or cervical surgery in the 2 years prior to inclusion.
* Patient participating in another clinical research protocol with an impact on the objectives of the research.
* Patient who is pregnant, breastfeeding or able to procreate without effective contraception*.
* Patient under guardianship, curatorship or deprived of liberty
* Patient under activated future protection mandate
* Patient under family habilitation
* Patient under court protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2027-09-25 (Estimated)

PRIMARY OUTCOMES:
Patients with a Neck Disability Index (NDI) score reduction of at least 7 points at M3. | At 3 months post cervical traction protocol
  The minimum clinically important difference (MCID) was established at 7 points out of 50 by (Cleland et al. 2006).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas RULLEAU, Principal Investigator — Nantes University Hospital
Locations (8):
- France (8):
  - CHD Vendée, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - CH Emile Roux, Le Puy-en-Velay
  - CHU Limoges, Limoges
  - CHU Nantes, Nantes
  - APHP La Pitié Salpêtrière, Paris
  - Chu Reims, Reims
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cormier G, Moreau C, Scalisi E, Pastor L, Rulleau T. The effect of mechanical traction on cervical radiculopathy: protocol for the TracCerv2 single-blind, randomised controlled trial. BMC Complement Med Ther. 2025 Feb 14;25(1):56. doi: 10.1186/s12906-025-04801-5. PMID 39953437